CLINICAL TRIAL: NCT06219187
Title: Male breAsT cAncer preDisposition Factor
Acronym: MATADOR
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 23 SEIN 02
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; PreDisposition factor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male breast cancer
  Interventions: Other: Questionnaire completion

INTERVENTIONS:
Other: Questionnaire completion — To meet the study's objective, patients will be asked to complete a questionnaire characterizing their environmental and psychosocial context.
  The questionnaire is to be completed by the patients themselves, or by their trusted support person as recorded in their medical records (in the particular case of a deceased patient).
  It is estimated that the questionnaire will take around 30 minutes to complete.
  Data will also be collected from the medical records of included patients:
  * Demographics
  * Disease data

SUMMARY:
This is a non-interventional, prospective, single-center study designed to collect and describe environmental and psychosocial data from patients with a history of male breast cancer (MBC) referenced in the IUCT-O regional database.

The study will be conducted on a population of 110 to 150 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male patient with a personal history of breast cancer
2. Age ≥ 18 years
3. Patient who has had an oncogenetic consultation at IUCT-O and is registered in the IUCT-O oncogenetic database
4. Patient for whom no pathogenic variant has been detected on the HBOC panel (HBOC-)
5. Patient with no objection to participation in the trial (for deceased patients: trusted support person with no objection to participation).

Exclusion Criteria:

1. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of male breast cancer (MBC) referenced in the IUCT-O's regional MutaFamily-MBC database.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
The environmental data in the questionnaire will be described by the usual descriptive statistics. | 15 days for each patient
  A 75-question questionnaire will cover such aspects as the patient's living conditions, professional situation, qualifications or level of education, social environment, early life and family environment, general health and recent significant events.
  Quantitative data will be described by the median, minimum, maximum and number of missing data, and qualitative data by the numbers, percentages and number of missing data for each modality.
Psychosocial data from the questionnaire will be described using standard descriptive statistics. | 15 days for each patient
  A 75-question questionnaire will cover such aspects as the patient's living conditions, professional situation, qualifications or level of education, social environment, early life and family environment, general health and recent significant events.
  Quantitative data will be described by the median, minimum, maximum and number of missing data, and qualitative data by the numbers, percentages and number of missing data for each modality.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France